CLINICAL TRIAL: NCT03572166
Title: Use of Copeptin Measurement After Arginine Infusion for the Differential Diagnosis of Diabetes Insipidus - the CARGOx Study
Acronym: CARGOx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University Hospital, Zürich (Other); Wuerzburg University Hospital (Other); Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other); Erasmus Medical Center (Other); Cambridge University Hospitals NHS Foundation Trust (Other); Federal University of Minas Gerais (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: CARGOx
Record Dates: First submitted 2018-06-04; First posted 2018-06-28 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Diabetes Insipidus; Polydipsia, Primary
Keywords: Copeptin
MeSH Terms: conditions — Diabetes Insipidus; Polydipsia, Psychogenic

STUDY DESIGN:
Intervention Model Description: Observational randomized cross-over diagnostic international multicenter study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arginine Infusion (Experimental): Arginine Stimulation Test
  Interventions: Diagnostic Test: Arginine infusion
- Hypertonic saline infusion (Active Comparator): Hypertonic Saline Infusion Test
  Interventions: Diagnostic Test: Hypertonic saline infusion

INTERVENTIONS:
Diagnostic Test: Arginine infusion — Intravenous Infusion of Arginine is given, copeptin measurement will be collected before and 60minutes after start of infusion
  Arms: Arginine Infusion
Diagnostic Test: Hypertonic saline infusion — Intravenous Infusion of hypertonic Saline is given, copeptin measurement will be collected before and once Plasma sodium rises above 149mmol/l
  Arms: Hypertonic saline infusion

SUMMARY:
The differential diagnosis of central diabetes insipidus (cDI) is difficult and the current test with the highest diagnostic accuracy is copeptin measurement after hypertonic saline infusion (HIS). Although the HIS improved diagnostic accuracy compared to the standard water deprivation test used for decades before, it still comprises great discomfort for patients due to the rise in serum sodium levels above 149mmol/l and requires the presence of medical staff at all times to guarantee safety of the test.

The arginine stimulation test is routinely used to stimulate growth hormone. Own data in 52 patients with polyuria / polydipsia syndrome showed that arginine infusion is a potent stimulator of the neurohypophysis and provides a new diagnostic tool in the differential diagnosis of cDI. Copeptin measurements upon arginine stimulation (CAS) discriminated patients with diabetes insipidus vs. patients with primary polydipsia with a high diagnostic accuracy of 94%.

To validate these results and to compare them against the HIS a large multicenter trial is needed, where the diagnostic accuracy of the CAS is compared to the HIS.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Hypotonic polyuria / polydipsia syndrome defined as: polyuria >50ml/kg body weight/24h and polydipsia >3l /24h or known diabetes insipidus under treatment with DDAVP
* Urine-Osmolality <800mOsm/L

Exclusion Criteria:

* Polyuria / polydipsia secondary to diabetes mellitus, hypercalcemia or hypokalemia
* Nephrogenic diabetes insipidus (defined as baseline copeptin level >21.4pmol/L)
* Evidence of any acute illness
* Epilepsy requiring treatment
* Uncontrolled arterial hypertension (blood pressure >160/100mmHg at baseline)
* Cardiac failure (NYHA III-IV)
* Liver cirrhosis (Child B-C)
* Uncorrected adrenal or thyroidal deficiency
* Patients refusing or unable to give written informed consent
* Pregnancy or breast feeding
* End of life care

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the overall diagnostic accuracy - defined as the proportion of correct diagnoses - of each diagnostic procedure in differentiating patients with central diabetes insipidus from patients with primary polydipsia. | 2 days
  For Arginine stimulation the copeptin cut-off to differentiate between diabetes insipidus and primary polydipsia will be 3.8 pmol/l after 60 minutes, for hypertonic saline stimulation it will be the copeptin cut-off 4.9 pmol/l taken at the end of the test

SECONDARY OUTCOMES:
Sensitivity of both diagnostic procedures for each diagnosis (Primary polydipsia, partial and complete central Diabetes insipidus) according to recommended diagnostic test criteria and previously generated cutoff values | 2 days (1 day for each test, evaluation diagnostic accuracy at end of trial)
  Copeptin cut-offs used:
  Arginine stimulation:
  * Copeptin level at 60 minutes < 2.4 pmol/l = complete central diabetes insipidus
  * Copeptin level at 60 minutes 2.4 - 3.8 pmol/l = partial central diabetes insipidus
  * Copeptin level at 60 minutes > 3.8 pmol/l = primary polydipsia
  Hypertonic saline stimulation:
  * Copeptin level < 2.7 pmol/l = complete central diabetes insipidus
  * Copeptin level 2.7 - 4.9 pmol/l = partial central diabetes insipidus
  * Copeptin level > 4.9 pmol/l = primary polydipsia
Specificity of both diagnostic procedures for each diagnosis (Primary polydipsia, partial and complete central Diabetes insipidus) according to recommended diagnostic test criteria and previously generated cutoff values | 2 days (1 day for each test, evaluation diagnostic accuracy at end of trial)
  Copeptin cut-offs used:
  Arginine stimulation:
  * Copeptin level at 60 minutes < 2.4 pmol/l = complete central diabetes insipidus
  * Copeptin level at 60 minutes 2.4 - 3.8 pmol/l = partial central diabetes insipidus
  * Copeptin level at 60 minutes > 3.8 pmol/l = primary polydipsia
  Hypertonic saline stimulation:
  * Copeptin level < 2.7 pmol/l = complete central diabetes insipidus
  * Copeptin level 2.7 - 4.9 pmol/l = partial central diabetes insipidus
  * Copeptin level > 4.9 pmol/l = primary polydipsia
Positive predictive value of both diagnostic procedures for each diagnosis (Primary polydipsia, partial and complete central Diabetes insipidus) according to recommended diagnostic test criteria and previously generated cutoff values | 2 days (1 day for each test, evaluation diagnostic accuracy at end of trial)
  Copeptin cut-offs used:
  Arginine stimulation:
  * Copeptin level at 60 minutes < 2.4 pmol/l = complete central diabetes insipidus
  * Copeptin level at 60 minutes 2.4 - 3.8 pmol/l = partial central diabetes insipidus
  * Copeptin level at 60 minutes > 3.8 pmol/l = primary polydipsia
  Hypertonic saline stimulation:
  * Copeptin level < 2.7 pmol/l = complete central diabetes insipidus
  * Copeptin level 2.7 - 4.9 pmol/l = partial central diabetes insipidus
  * Copeptin level > 4.9 pmol/l = primary polydipsia
Negative predictive value of both diagnostic procedures for each diagnosis (Primary polydipsia, partial and complete central Diabetes insipidus) according to recommended diagnostic test criteria and previously generated cutoff values | 2 days (1 day for each test, evaluation diagnostic accuracy at end of trial)
  Copeptin cut-offs used:
  Arginine stimulation:
  * Copeptin level at 60 minutes < 2.4 pmol/l = complete central diabetes insipidus
  * Copeptin level at 60 minutes 2.4 - 3.8 pmol/l = partial central diabetes insipidus
  * Copeptin level at 60 minutes > 3.8 pmol/l = primary polydipsia
  Hypertonic saline stimulation:
  * Copeptin level < 2.7 pmol/l = complete central diabetes insipidus
  * Copeptin level 2.7 - 4.9 pmol/l = partial central diabetes insipidus
  * Copeptin level > 4.9 pmol/l = primary polydipsia
Best fit diagnostic copeptin cut-off values for differentiation between each diagnosis (Primary polydipsia, partial and complete central Diabetes insipidus) upon arginine stimulation and hypertonic saline infusion stimulation | 2 days (1 day for each test, evaluation diagnostic accuracy at end of trial)
Accuracy of the copeptin cut-off of 3.7 pmol/l after 60 minutes and 4.1 after 90 minutes for Arginine Stimulation test | 2 days (1 day for each test, evaluation diagnostic accuracy at end of trial)
Sensitivity of the copeptin cut-off of 3.7 pmol/l after 60 minutes and 4.1 after 90 minutes for Arginine Stimulation test | 2 days (1 day for each test, evaluation diagnostic accuracy at end of trial)
Specificity of the copeptin cut-off of 3.7 pmol/l after 60 minutes and 4.1 after 90 minutes for Arginine Stimulation test | 2 days (1 day for each test, evaluation diagnostic accuracy at end of trial)
Accuracy of the copeptin cut-off of 6.5 pmol/l for Hypertonic Saline Infusion test | 2 days (1 day for each test, evaluation diagnostic accuracy at end of trial)
Sensitivity of the copeptin cut-off of 6.5 pmol/l for Hypertonic Saline Infusion test | 2 days (1 day for each test, evaluation diagnostic accuracy at end of trial)
Specificity of the copeptin cut-off of 6.5 pmol/l for Hypertonic Saline Infusion test | 2 days (1 day for each test, evaluation diagnostic accuracy at end of trial)
Frequency and severity of thirst assessed by visual analogue scale during both tests | 2 days (1 for each test)
  assessed by visual analogue scale from 0 to 10, with 0 indicating no symptoms and 10 indicating severe symptoms.
Frequency and severity of headache assessed by visual analogue scale during both tests | 2 days (1 for each test)
  assessed by visual analogue scale from 0 to 10, with 0 indicating no symptoms and 10 indicating severe symptoms.
Frequency and severity of nausea assessed by visual analogue scale during both tests | 2 days (1 for each test)
  assessed by visual analogue scale from 0 to 10, with 0 indicating no symptoms and 10 indicating severe symptoms.
Frequency and severity of vertigo assessed by visual analogue scale during both tests | 2 days (1 for each test)
  assessed by visual analogue scale from 0 to 10, with 0 indicating no symptoms and 10 indicating severe symptoms.
Frequency and severity of general malaise assessed by visual analogue scale during both tests | 2 days (1 for each test)
  assessed by visual analogue scale from 0 to 10, with 0 indicating no symptoms and 10 indicating severe symptoms.
Subjective burden assessed by visual analogue scale of both tests | 2 days (1 for each test)
  assessed by visual analogue scale from 0 to 10, with 0 indicating no symptoms and 10 indicating severe symptoms.
Health care costs of both tests | 2 days (1 for each test)
Frequency of test preference at follow up visit | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam Christ-Crain, Prof, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (7):
- Hospital das clinicas Minas Gerais, Belo Horizonte, Brazil
- University Hospital Würzburg, Würzburg, Germany
- Granda Ospedale Maggiore Policlinico Milan, Milan, Italy
- Erasmus MC, Rotterdam, Netherlands
- Switzerland (2):
  - University Hospital Basel, Department of Endocrinology, Basel, Canton of Basel-City
  - University Hospital Zurich, Zurich
- Cambridge University Hospital, Cambridge, United Kingdom

REFERENCES:
- [Derived] Atila C, Chifu I, Drummond JB, Vogt DR, Nahum U, Fassnacht M, Winzeler B, Refardt J, Christ-Crain M. A novel diagnostic score for diagnosing arginine vasopressin deficiency (central diabetes insipidus) or primary polydipsia with basal laboratory and clinical parameters: results from two international multicentre prospective diagnostic studies. Lancet Diabetes Endocrinol. 2025 Jun;13(6):505-515. doi: 10.1016/S2213-8587(25)00053-1. Epub 2025 Apr 25. PMID 40294614
- [Derived] Bizzozero CA, Monnerat S, Chapman FA, Dhaun N, Refardt J, Christ-Crain M. Apelin levels in patients with polyuria-polydipsia syndrome upon copeptin stimulation tests. Eur J Endocrinol. 2024 Oct 29;191(5):491-498. doi: 10.1093/ejendo/lvae138. PMID 39425917
- [Derived] Refardt J, Atila C, Chifu I, Ferrante E, Erlic Z, Drummond JB, Indirli R, Drexhage RC, Sailer CO, Widmer A, Felder S, Powlson AS, Hutter N, Vogt DR, Gurnell M, Soares BS, Hofland J, Beuschlein F, Fassnacht M, Winzeler B, Christ-Crain M. Arginine or Hypertonic Saline-Stimulated Copeptin to Diagnose AVP Deficiency. N Engl J Med. 2023 Nov 16;389(20):1877-1887. doi: 10.1056/NEJMoa2306263. PMID 37966286